CLINICAL TRIAL: NCT04812067
Title: A Phase 2 Clinical Trial to Assess the Safety and Observe the Potential Benefit of TTHX1114 Delivered Via Intra-Cameral (IC) Injection
Brief Title: A Safety and Efficacy Trial of TTHX1114 in People With CED
Acronym: OPTIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trefoil Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTHX-901
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Corneal Endothelial Dystrophy
MeSH Terms: conditions — Corneal Dystrophy, Posterior Polymorphous, 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TTHX1114 weekly x 5 (Experimental): TTHX1114 via IC injection weekly x 5
  Interventions: Drug: TTHX1114

INTERVENTIONS:
Drug: TTHX1114 — engineered FGF-1

SUMMARY:
Expanded access, open label study at a single dose level in patients with CED that in the opinion of the investigators might benefit from TTHX1114

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older
* Subjects who are women of childbearing potential (WOCBP) must be using an acceptable method of birth control (See Section 6.4.3)
* Proposed Study Eye that has been diagnosed with an ocular condition that, in the opinion of the Investigator, could possibly benefit from TTHX1114 administration, and has a measurable efficacy endpoint
* Fellow Eye with 20/100 BCVA or better
* No concurrent ocular or medical condition that would impair the assessment of safety and efficacy

Exclusion Criteria:

* Prior exposure to TTHX1114
* Intolerance, hypersensitivity, or significant allergy to any drug compound, food, or other substance (Note: This includes all components and excipients of the study drug)
* Current or recent (e.g., the 28 days prior to Study Day 0) participation in any other, interventional clinical research study
* History of:

  * Ocular cancer (including melanoma)
  * Herpetic keratitis
  * Documented and repeated elevated IOP in either eye
  * Posterior Polymorphous Corneal Dystrophy (PPCD; aka Schlichting dystrophy)
  * Uveitis
* Use of any concomitant medications that may interfere with the assessment of safety and efficacy
* Any other reason (e.g., serious systemic disease or uncontrolled medical condition) that, in the opinion of the Investigator could increase the subject's risk, interfere with the interpretation of the study results, or affect the subject's ability to provide informed consent or comply with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Specular Microscopy | Day 28
  Corneal Endothelial Cell Density

SECONDARY OUTCOMES:
Pachymetry | Day 28
  Central Corneal Thickness

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Tremblay, Study Director — Trefoil Therapeutics.com
Locations (2):
- United States (2):
  - Trefoil Study Site, Atlanta, Georgia
  - Trefoil Study Site, Washington, Missouri

IPD SHARING:
Plan to Share IPD: No